CLINICAL TRIAL: NCT01108393
Title: Efficacy of Agomelatine 25mg/Day (With Possible Increase to 50mg/Day After 8 Weeks of Treatment) Given Orally During 16 Weeks in Patients With Obsessive-Compulsive Disorder. A Randomised, Double-blind, Placebo-controlled, Parallel Groups, International Study
Brief Title: Efficacy of Agomelatine in Patients With Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL2-20098-072; 2009-016713-20 (EudraCT Number)
Record Dates: First submitted 2010-04-09; First posted 2010-04-22 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2020-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Agomelatine
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Agomelatine A (Experimental)
  Interventions: Drug: Agomelatine A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Agomelatine A — Agomelatine 25 mg film-coated tablet
  Agomelatine 2x25mg film-coated tablet
  Arms: Agomelatine A
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy of agomelatine compared to placebo on the reduction of Obsessive and Compulsive symptoms after 16 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Obsessive Compulsive Disorder (OCD) according to Diagnostic and Statistical Manual, Fourth Edition, Text Revision (DSM-IV-TR),
* Y-BOCS total score ≥ 20,
* duration of OCD symptoms of at least one year.

Exclusion Criteria:

* Bipolar disorder, Schizophrenic or Psychotic Disorder
* Severe or uncontrolled organic diseases
* Neurological disorder
* Women of childbearing potential who are not using effective contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Y-BOCS total score | 16 weeks
  Yale-Brown Obsessive Compulsive scale (Y-BOCS) total score. This scale measures the severity of obsessive and compulsive symptoms from baseline to W16.

SECONDARY OUTCOMES:
NIMH-OC score | 16 weeks
  National Institute for Mental Health- Obsessive Compulsive scale (NIMH-OC) Total Score. This scale measures the severity of obsessive and compulsive symptoms from baseline to week 16.
MADRS total score | 16 weeks
  Montgomery and Asberg Depression rating scale (MADRS) Total score. This scale measures the severity of depressive symptoms from baseline to week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, Prof., Principal Investigator — Department of Psychiatry Chaim Sheba Medical Center
Locations (1):
- Department of Psychiatry Chaim Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies in patients:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com